CLINICAL TRIAL: NCT03816306
Title: Six Months Clinical and Echocardiographic Outcome of Angiotensin Receptor-Neprilysin Inhibitor (ARNI) LCZ696 Therapy in Heart Failure Patients With Reduced Ejection Fraction (HFrEF)
Brief Title: Six Months Clinical and Echocardiographic Outcome of ARNI LCZ696 Therapy in HFrEF Patients
Status: Completed | Type: Observational
Sponsor: Mohammed Alnims (Other)
Responsible Party: Sponsor-Investigator, Mohammed Alnims, Doctor, Investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 31640
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single group study
  Interventions: Drug: LCZ 696

INTERVENTIONS:
Drug: LCZ 696 — LCZ696 is an Angiotensin receptor neprilysin inhibitor. It's composed of Sacubitril/Valsartan. LCZ696 starting dose 50 mg P.O. BID, LCZ696 100 mg P.O. BID and up-titration to LCZ696 200 mg P.O. BID.

SUMMARY:
To evaluate the clinical and echocardiographic outcome of LCZ696 therapy in HFrEF (NYHA Class II - IV and EF =≤ 40%).patients, in addition to the efficacy of LCZ696 in reducing mortality and rehospitalisation rate.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 year old.
2. Functional class using New York Heart Association (NYHA) classification class II, III or IV %).
3. Left ventricular systolic dysfunction using transthoracic echocardiography with EF ≤ 40%.
4. Who was already taking ACE inhibitors or ARBs.

Exclusion Criteria:

1. Symptomatic hypotension.
2. Systolic blood pressure <100 mm Hg.
3. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2.
4. History of angioedema.
5. Hisotry of unacceptable side effects while on while on treatment with an ACE-inhibitor or ARBs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any Patients with HFrEF (EF ≤ 40%) above 18 year old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants That Had Either Cardiovascular (CV) Death or Heart Failure (HF) Hospitalization. | 6 Months after starting LCZ696 Therapy
  Number of participants that had either CV death or HF hospitalization due to HF.
Change From Baseline to Month 6 for The Minnesota Living with Heart Failure Questionnaire (MLHFQ). | 6 Months after starting LCZ696 Therapy
  Change From Baseline to Month 6 for the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The questionnaire was designed as a self-administered measure of the effects of heart failure and treatments for heart failure on patients' quality of life. The questionnaire has 21 items assess the impact of frequent physical symptoms of heart failure and the effects of heart failure on physical and social functions. The response scale for all 21 items on the MLHF is based on a 6-point ( from 0 to 5 ). Scores are transformed to a range of 0-105, in which higher scores reflect better health status.

SECONDARY OUTCOMES:
Number of Patients - All-cause Mortality. | 6 Months after starting LCZ696 Therapy
  Number of patients - All-cause mortality. All-cause mortality is common in HF patients.
Number of Patients With First Confirmed Renal Dysfunction. | 6 Months after starting LCZ696 Therapy
  Number of patients with first confirmed renal dysfunction ( a decrease in the eGFR of at least 50% or a decrease of more than 30 ml per minute per 1.73 m2 to less than 60 ml per minute per 1.73 m2 ).
Number of Patients with Changes in The Left Ventricular Systolic Function (EF). | 6 Months after starting LCZ696 Therapy
  Number of Patients with improvement in the ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Abdelhamid, MD, FACC, FESC, FSCAI, Study Director — Professor of Cardiovascular Medicine, Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No